CLINICAL TRIAL: NCT02365909
Title: A Prospective Randomized Double-Blind Placebo Controlled Study Evaluating Sphenopalatine Ganglion Block (SPGB) for Treatment of Postdural Puncture Headache (PDPH)
Brief Title: Study Evaluating Sphenopalatine Ganglion Block (SPGB) for Treatment of Postdural Puncture Headache (PDPH)
Acronym: PDPH
Status: Terminated | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Study stopped due to difficulty recruiting patients
Sponsor: University of Arkansas (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 203684
Record Dates: First submitted 2015-02-11; First posted 2015-02-19 (Estimated); Last update posted 2017-09-18 (Actual); Status verified 2017-09

CONDITIONS: Postdural Puncture Headache
MeSH Terms: conditions — Post-Dural Puncture Headache | interventions — Bupivacaine; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Acitve (Active Comparator): This group will receive 0.3 ml of 0.5% bupivacaine per nare, applied with the Tx360®
  Interventions: Drug: 0.5% bupivacaine
- Placebo (Placebo Comparator): This group will receive 0.3 ml of normal saline per nare, applied with the Tx360®
  Interventions: Drug: normal saline

INTERVENTIONS:
Drug: 0.5% bupivacaine — This group will receive 0.3 ml of 0.5% bupivacaine per nare, applied with the Tx360®
  Arms: Acitve
Drug: normal saline — This group will receive 0.3 ml of normal saline per nare, applied with the Tx360®
  Arms: Placebo

SUMMARY:
Postdural puncture headaches (PDPH) are a consequence of spinal and epidural anesthesia in approximately 1% of cases when performed in obstetric patients. The gold standard treatment for a PDPH is currently an epidural blood patch (EBP), which involves placing a needle back into the epidural space of the neuraxium and then injecting 20 ml of the patient's own blood through the needle and into the epidural space to form a clot over the insult in the tissue layer that causes the headaches. The investigators want to test the efficacy of using a less invasive procedure, called a sphenopalatine block (SPGB), for treatment of PDPH. SPGB has been used for many years in the treatment of migraines and cluster headaches, and there are several case reports of its use to successfully treat PDPH as well. SPGB simply involves applying a local anesthetic to the mucosa in the back of each nostril to numb the nerves that cause the headache. The investigators hope that the SPGB will reduce the number of PDPH patients that require and EBP.

ELIGIBILITY:
Inclusion Criteria

* Active postdural puncture headache within 7 days after neuraxial analgesia/anesthesia
* Age ≥ 18 years.
* ASA physical status ≤ 3

Exclusion Criteria

* Known coagulopathy
* Known nasal septal deviation or abnormalities
* Medical conditions contraindicated to bupivacaine or the nasal applicator (according to the product labeling)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2015-06-29 (Actual); Primary Completion 2016-08-30 (Actual); Study Completion 2016-08-30 (Actual)

PRIMARY OUTCOMES:
Headache verbal pain score | 1 hour

CONTACTS AND LOCATIONS:
Locations (1):
- University of Arkansas for Medical Sciences, Little Rock, Arkansas, United States